CLINICAL TRIAL: NCT06071572
Title: San Raffaele IBD Biobank: Accelerating Research From the Bed to the Bench Side
Brief Title: San Raffaele IBD Biobank
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvio Danese, Director of Gastroenterology and Endoscopy Unit, IRCCS San Raffaele
Other Study IDs: IBD Biobank
Record Dates: First submitted 2023-09-25; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biological samples collected specifically for the IBD Biobank — Biological samples will include: material intestinal biological waste (surgical leftover), 30 ml of peripheral blood, one sample stool standards and a saliva sample.

SUMMARY:
The developments of knowledge and possibilities of investigation in the biomedical field, and in particularly in the field of inflammatory bowel diseases need to be analyzed and study vast cases of biological material carefully collected, preserved and correlated with complete clinical-pathological-instrumental data. In order to organize and make uniform the collection, storage and management of samples and the clinical data associated with them, a biobank is being set up, called "IBD Biobank" aimed at studying inflammatory intestinal diseases. THE subjects/patients who decide to authorize the collection, storage and use of biological material for future research purposes which are not currently identifiable will be called, in this document, donors. The IBD Biobank involves the recruitment of adult subjects. To each donor will be given informed consent DSAN 1178/6 ("Regulation e informed consent for the collection, conservation and use of human biological material spontaneous monocentric or multicentric studies with promoting OSR") or the most updated version of this informed consent, according to the directives of the OSR Ethics Committee. The biological material of the IBD Biobank will be processed at the laboratories of the Biological Resources Center (CRB) e preserved at BIOREP srl (Via Olgettina, 60, c/o San Raffaele Hospital-DIBIT2 - Palazzina San Michele 20132 Milan). Generally biological materials will be collected during the already scheduled surgery and the routine clinical examination as part of outpatient visits, day hospitals and hospital admissions. The biological samples will come stored in tubes equipped with barcode identification (2D) which guarantee a code unique to each rate and preserve its anonymity. The clinical-pathological-instrumental data, demographic and anamnestic information will be entered by trained personnel on a computerized database anonymously by assigning a UPN code identifying the patient. Access the database is managed via personal login and password. All data entered is recorded and stored on the server of the IRCCS San Raffaele Hospital in Milan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBD (min 18 years)

Exclusion Criteria:

* Patients without IBD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll Patients with IBD affering to OSR
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-01-18 (Estimated); Study Completion 2026-01-18 (Estimated)

PRIMARY OUTCOMES:
To perform DNA, RNA and protein extraction, cell isolation, serum isolation and metabolomic analysis from IBD patients blood, tissue, feces and saliva | 1-36
  In particular, the analysis are:
  Tissue: DNA, RNA and protein extraction, cell isolation Blood: DNA, RNA and protein extraction, cell isolation and serum isolation Feces: DNA and RNA extraction, metabolomic analysis Saliva: DNA and RNA extraction

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided